CLINICAL TRIAL: NCT02218307
Title: The Use of Antibiotic Sinonasal Rinse After Sinus Surgery: A Randomized Double-Blind Control Trial
Brief Title: The Use of Antibiotic Sinonasal Rinse After Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Roy R. Casiano, Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20110846
Record Dates: First submitted 2014-07-10; First posted 2014-08-18 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Chronic Rhinosinusitis
MeSH Terms: interventions — Mupirocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mupirocin (Active Comparator): topical antibiotic
  Interventions: Drug: Mupirocin
- Placebo (Placebo Comparator): Placebo control for mupirocin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mupirocin
  Arms: Mupirocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Double blind placebo controlled trial to evaluate whether the routine use of nasal irrigation with mupirocin is more effective than saline irrigations alone in reducing symptoms of chronic rhinosinusitis in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Rhinosinusitis
* Undergoing endoscopic sinus surgery

Exclusion Criteria:

* Age under 18
* Documented adverse reaction to mupirocin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Miller School of Medicine, ENT Dept, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mupirocin: topical antibiotic
  Mupirocin
- Placebo: Placebo control for mupirocin
  Placebo
Period: Overall Study
Arm/Group | Mupirocin | Placebo
Started | 34 | 34
Completed | 25 | 33
Not Completed | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mupirocin | Placebo | Total
Number analyzed (Participants) | 25 | 33 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 26 | 46
  >=65 years | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life in Chronic Rhinosinusitis Patients
Description: Measuring the quality of life in chronic rhinosinusitis through completion of a questionnaire named SNOT 20 ( 20 questions for Sino-Nasal Outcome Test)
  Snot20:
  Scale 1 to 5 for 20 symptoms numbered below where 5 is the worst symptom. Total SNOT is scale from 0-100 where 100 is the worst.
  The following are the elements:
  1. need to blow 2. sneezing 3. runny nose 4. cough 5. postnasal drip 6. Thick nasal discharge 7. Ear fullness 8. Dizziness 9. Ear pain 10. facial pain/pressure 11. difficulty falling asleep 12. wake up at night 13. lack of a good night's sleep 14. wake up tired 15. Fatigue 16. Reduced productivity 17. Reduced concentration 18. frustrated/ restless/irritable 19. sad 20. Embarrassed
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Mupirocin | Placebo
Number analyzed (Participants) | 24 | 32
Units on a scale | 23 (19.23) | 21 (17.33)

2. Secondary Outcome: Quality of Life in Chronic Rhinosinusitis Patients
Description: Measuring the quality of life in chronic rhinosinusitis through completion of a questionnaire named Visual Analog Scale for Nasal Obstruction/Congestion. VAS for nasal obstruction is scale from 0 to 100 where 100 mean worse.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Mupirocin | Placebo
Number analyzed (Participants) | 25 | 33
Units on a scale | 24.8 (25.64) | 26.4 (26.13)

ADVERSE EVENTS:
Arm/Group | Mupirocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/33
Other Adverse Events (participants affected / at risk) | 0/25 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes